CLINICAL TRIAL: NCT01353586
Title: REVOLUTION (WFCC-133): Clinical Workflow Study for the Evaluation of the Multi-Electrode Pulmonary Vein Isolation System for the Treatment of Paroxysmal Atrial Fibrillation (PAF)
Brief Title: REVOLUTION (WFCC-133) - Treatment of Paroxysmal Atrial Fibrillation
Acronym: REVOLUTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WFCC-133
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radionuclide Generators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- nMARQ™ System (Experimental): The nMARQ™ System (Circular and Crescent Mapping and Ablation Catheters as well as the Multi-Channel Radiofrequency Generator) as part of the Multi-Electrode Irrigated Pulmonary Vein (PV) Isolation System will serve as a treatment method for subjects undergoing radiofrequency catheter ablation for drug refractory, symptomatic Paroxysmal Atrial Fibrillation (PAF). The study later included a Subpopulation Neurological Assessments (SNA) substudy which is a prospective, non-randomized, controlled, acute assessment to compare subjects treated with the nMARQ™ System against control subjects treated with the NAVISTAR® THERMOCOOL® Irrigated Tip Catheter.
  Interventions: Device: nMARQ™ System

INTERVENTIONS:
Device: nMARQ™ System — The nMARQ™ System is indicated for catheter-based electrophysiological mapping for the treatment of drug refractory recurrent symptomatic paroxysmal atrial fibrillatioon.
  Other Names: nMARQ™ Circular and Crescent Mapping and Ablation Catheters; Circular/Crescent Ablation Catheters; nMARQ™ Catheters; Circular/Crescent Irrigated catheters; Multi-Channel Radiofrequency (RF) Generator; nMARQ™ Generator; nMARQ™ Multi-Electrode Irrigated Pulmonary Vein (PV)

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the Circular and Crescent Mapping and Ablation catheters and the workflow of the Multi-Electrode Irrigated Pulmonary Vein Isolation System when used for the treatment of drug refractory symptomatic paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
The study will include a Workflow Phase to verify consistent workflow of all study device components and evaluate acute safety. Upon meeting the defined criteria, the Workflow Phase will be closed and further enrollment will be toward the Main Study Phase which includes the roll-in (the first 3 subjects enrolled at each site following the closure of the Workflow Phase) and Subpopulation Neurological Assessments (SNA) substudy subjects. SNA assessment is a prospective, non-randomized, controlled, acute assessment of two ablation devices to determine if intracerebral microemboli are generated during or immediately after radiofrequency ablation therapy for PAF. SNA subjects will remain and complete the Main Study Phase. However, SNA-control subjects will not be considered part of the Main Study Phase. All subjects, including the subjects enrolled under the Workflow Phase will be included in the Safety Cohort (evaluated for Primary Safety endpoint and all Secondary Safety endpoints).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic Paroxysmal Atrial Fibrillation (PAF) who have had at least one documented Atrial Fibrillation (AF) episode in the twelve (12) months prior to enrollment. Documentation may include electrocardiogram (ECG), transtelephonic monitor (TTM), Holter Monitor (HM), or telemetry strip.
2. Failure of at least one antiarrhythmic drug for AF (class I or III, or Atrioventricular (AV) nodal blocking agents such as beta blockers and calcium channel blockers), as evidenced by recurrent symptomatic AF, or intolerable side effects.
3. Age 18 years or older.
4. Able and willing to comply with all pre-, post- and follow-up testing and requirements.
5. Signed Patient Informed Consent Form.

Exclusion Criteria:

1. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
2. Patients with Persistent or Long-standing AF (AF episode lasting > 30 days in duration.
3. Diagnosed atrial myxoma.
4. Left atrial size > 5.5cm.
5. Left Ventricular ejection fraction < 40%.
6. Contraindication to Computed Axial Tomography/Magnetic Resonance Imaging (CT/MRI) procedures
7. New York Heart Association Class III or IV.
8. Previous ablation for enrolled arrhythmia (AF).
9. Documented left atrial thrombus on imaging (example: transesophageal echocardiography or intracardiac echocardiography).
10. Myocardial Infarction within the previous 60 days (2 months).
11. Any valvular cardiac surgical procedure (that is, valve repair or replacement and presence of a prosthetic valve).
12. Coronary artery bypass graft procedure with the last 180 days 6 months.
13. Cardiac Surgery (that is, ventriculotomy, atriotomy) within the past 60 days (2 months).
14. Awaiting cardiac transplantation or other cardiac surgery within the next 365 days (12 months).
15. History of documented thromboembolic event within the past one (1) year.
16. Significant pulmonary disease, (example: restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunctions of the lungs or respiratory system that produces chronic symptoms.
17. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
18. Active illness or active systemic infection or sepsis.
19. Unstable angina.
20. History of blood clotting or bleeding abnormalities.
21. Contraindication to anticoagulation (that is, Heparin or Warfarin).
22. Life expectancy less than 365 days (12 months)
23. Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation.
24. Women who are pregnant (as evidence by pregnancy test if subject is of child bearing potential) and/or breast feeding.
25. Presence of a condition that precludes vascular access.
26. Enrollment in an investigational study evaluating another device or drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2013-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Pierre Jais, MD, Principal Investigator — Hop. Haut-Lévêque
Locations (8):
- AZ St Jan, Cardiologie, Bruges, Belgium
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia
- HCV HjerteCenter Varde, Varde, Denmark
- France (2):
  - HHL Hop. Haut-Lévêque, Bordeaux
  - HDB CHU de Nancy, Nancy
- HLG Herzzentrum Leipzig GmbH, Leipzig, Germany
- Italy (2):
  - OFM Ospedale Generale Regionale, Acquaviva delle Fonti
  - CCM Centro Cardiologico Monzino, Milan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 186 eligible subjects enrolled in this study across 8 sites in Europe. The first was enrolled on March 14, 2011 and was treated on March 15, 2011. The last was enrolled on October 16, 2012. The study's last 12 month follow-up visit occurred on September 27, 2013.
Pre-assignment Details: The Main Study consisted only of subjects treated with nMARQ ablation system, without a control arm. Later, a Subpopulation Neurological Assessment (SNA) was added to evaluate for potential cerebral micro-emboli and neurological deficits post ablation. The SNA included a comparator control arm of subjects treated with the Navistar® ThermoCool®.
Groups:
- nMARQ™ (Main Study- Single Arm): This group of subjects underwent electrophysiological mapping and radiofrequency ablation with the Biosense Webster nMARQ™ system. The Main Study (167 subjects) consists only of subjects treated with the nMARQ catheter.
- NAVISTAR® THERMOCOOL® (SNA Subpopulation Only): Version 3.0 of the Clinical Investigation Plan added a Subpopulation Neurological Assessments (SNA) designed to evaluate post-ablation generation of cerebral microemboli and associated neurological deficits.
  These assessments were done in a prospective, non-randomized manner, comparing subjects treated with the nMARQ system against control subjects treated with the NAVISTAR® THERMOCOOL® Irrigated Tip Catheter.
  Per study design, the data from the NAVISTAR® THERMOCOOL® subpopulation would be used for SNA analysis only. The data in this column are presented for transparency; but cannot be compared statistically against the data from the Main Study group.
Period: Overall Study
Arm/Group | nMARQ™ (Main Study- Single Arm) | NAVISTAR® THERMOCOOL® (SNA Subpopulation Only)
Started | 167 | 19
Participated in Workflow Phase | 20 | 0
Participated in Roll-in Phase | 22 | 0
Participated in SNA Substudy | 19 | 19
Completed | 160 | 17
Not Completed | 7 | 2
Not completed — Procedure terminated prior to ablation | 3 | 0
Not completed — Never had insertion of study catheter | 4 | 1
Not completed — Neurological exam not done | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population (cohort): For the main study, this population includes enrolled subjects who underwent insertion of study catheters. For the NAVISTAR® THERMOCOOL® arm, this population includes enrolled subjects, but excludes two subjects (1 with low pre-ablation international normalized ratio (INR) and 1 missing post procedure neurological exam).
Groups:
- Total: Total of all reporting groups
Arm/Group | nMARQ™ (Main Study- Single Arm) | NAVISTAR® THERMOCOOL® (SNA Subpopulation Only) | Total
Number analyzed (Participants) | 163 | 17 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.24) | 56.5 (9.86) | 58.49 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 3 | 54
  Male | 112 | 14 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 110 | 14 | 124
  Unknown or Not Reported | 53 | 3 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants] — Fifty-three subjects in nMARQ arm and 3 subjects in SNA Control Group didn't report ethnicity and race data because of French privacy law restrictions. These subjects are reported in Race category, "Unknown or Not Reported".
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 110 | 14 | 124
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 53 | 3 | 56

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Early Onset Primary Adverse Events
Description: The primary safety endpoint is the incidence of early onset primary adverse events within 7 days of the mapping and ablation procedure. Primary adverse events include pericardial effusion requiring intervention, atrial perforation, pericarditis requiring intervention, cardiac tamponade, pneumothorax, death, pulmonary edema, diaphragmatic paralysis, heart block, stroke / cerebrovascular accident (CVA), hospitalization (initial and prolonged), thromboembolism, myocardial infarction (MI), transient ischemic attack (TIA), and vascular access complications. In addition, pulmonary vein stenosis and atrio-esophageal fistula that occurs greater than one week (7 days) post-procedure are deemed primary adverse event.
Time Frame: Any of above events occurring within 7 days post-procedure (also including the incidence of pulmonary vein stenosis and atrio-esophageal fistula occurring > 7 days and up to one year post-procedure)
Population: Safety Population as defined above
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- nMARQ™ (Main Study- Single Arm): The Main Study group consists of subjects who were treated with the Biosense Webster nMARQ™ system. This group is single-arm and does not include the SNA substudy population (no comparator group).
Arm/Group | nMARQ™ (Main Study- Single Arm)
Number analyzed (Participants) | 163
percentage of participants | 5.5 [2.6 to 10.2]

2. Primary Outcome: Incidence of Freedom From Documented Symptomatic Atrial Fibrillation
Description: The primary effectiveness endpoint is freedom from documented symptomatic atrial fibrillation based on electrocardiographic data through 8 months post ablation.
Time Frame: Evaluated from Day 91 to Day 240
Population: Effectiveness cohort: This population excludes those subjects who never underwent insertion of study catheter, those who terminated procedure prior to ablation, and those who were enrolled during the Workflow phase (20 subjects) and Roll-in phase (22 subjects). This analysis also excludes two subjects who withdrew consent post ablation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | nMARQ™ (Main Study- Single Arm)
Number analyzed (Participants) | 116
percentage of participants | 71.6 [62.4 to 79.5]
Statistical Analysis 1: Comparison: nMARQ™ (Main Study- Single Arm); Test type: Superiority or Other; Proportion of events = 71.6, 95% CI 2-sided [63.3 to 79.8] — The above supplemental analysis is to estimate the rate of subjects without documented symptomatic AF at Day 240 using the Kaplan-Meier time-to-event analysis method to accommodate the censored information from the two withdrawn subjects

3. Secondary Outcome: Incidence of Non-Primary Serious Adverse Events (SAEs) up to 12 Months
Description: This secondary safety endpoint includes non-primary serious adverse events within 7 days post-procedure and serious adverse events from 7 days to 12 months post-procedure.
Time Frame: 12 months post study procedure
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | nMARQ™ (Main Study- Single Arm)
Number analyzed (Participants) | 163
percentage of participants
  Non-primary serious AEs within 7 days | 0.6
  Serious adverse events from 7 days to 12 months | 15.3

4. Secondary Outcome: Assessment of Pulmonary Vein (PV) Narrowing and Stenosis at 3 Months After Index Ablation
Description: Incidence of narrowing of PV and stenosis at 3 months post ablation, for subjects with available CT/MRA scans at 3 months. PV Stenosis is defined as 70% or more PV diameter reduction.
Time Frame: Three months after index ablation
Population: Subjects in safety analysis group who also had CT/MRI PV scan available at the 3-month post-ablation interval (144 of 160 subjects)
Measure: Number; unit: percentage of participants with CT/MRI
Groups:
- nMARQ™ System (Main Study - Single Arm): The Main Study group consists of subjects who were treated with the Biosense Webster nMARQ™ system. This group is single-arm and does not include the SNA substudy population (no comparator group).
Arm/Group | nMARQ™ System (Main Study - Single Arm)
Number analyzed (Participants) | 144
percentage of participants with CT/MRI
  0-20% Reduction of PV Diameter | 47.2
  21- 50% Reduction of PV Diameter (Mild) | 51.4
  51-70% Reduction of PV Diameter (Moderate) | 1.4
  > 70% Reduction of PV Diameter (Severe) | 0.0

5. Secondary Outcome: Incidence of Completion of Ablation Procedure
Description: This secondary outcome describes the acute effectiveness, which is defined as pulmonary vein isolation (PVI) documented by confirmed entrance block (with or without the use of a focal catheter).
Time Frame: From 7 days to 12 months post study procedure
Population: Safety population excluding one subject without source document at site
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | nMARQ™ System (Main Study - Single Arm)
Number analyzed (Participants) | 117
percentage of participants | 100 [96.9 to 100]

6. Secondary Outcome: Absence of Documented Symptomatic PAF Through 6 Months and 12 Months Post Procedure
Description: This endpoint is defined as the absence of documented symptomatic PAF recurrence through 6 months and 12 months post index ablation procedure.
Time Frame: 6 and12 months post study procedure
Population: This analysis population is the effectiveness cohort, excluding 2 subjects who withdrew consent prior to Day 91. The effectiveness cohort includes those who received treatment with the investigational device; but does not include 20 workflow and 22 roll-in subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | nMARQ™ System (Main Study - Single Arm)
Number analyzed (Participants) | 116
percentage of participants
  6 months post ablation | 73.3 [64.3 to 81.1]
  12 months post ablation | 60.3 [50.8 to 69.3]

7. Secondary Outcome: Subpopulation Neurological Assessments (SNA) Endpoint 1 - Incidence of Cerebral Embolic (ACE) Lesions Post Ablation
Description: Evaluation of post-ablation generation incidence of asymptomatic cerebral microembolic lesions post ablation, as documented by MRI. All microembolic lesions reported in this study are asymptomatic.
Time Frame: 48 hours post-ablation
Population: Neurological assessment subpopulation. This population includes 19 subjects from the nMARQ main study and 17 subjects from the Thermocool control group.
Measure: Number; unit: percentage of subjects with ACE Lesion
Groups:
- nMARQ™ System (SNA Subpopulation): The nMARQ arm of the SNA subpopulation included 19 subjects treated with the nMARQ™ System.
Arm/Group | nMARQ™ System (SNA Subpopulation) | NAVISTAR® THERMOCOOL® (SNA Subpopulation Only)
Number analyzed (Participants) | 19 | 17
percentage of subjects with ACE Lesion | 21.1 | 5.9

8. Secondary Outcome: Subpopulation Neurological Assessments (SNA) Endpoint 2 - Incidence of New Neurological Findings Post Ablation
Description: All SNA subjects were to be evaluated by expert neurologists for existing neurological deficits prior to ablation procedure. After procedure, those subjects were also to be assessed for new neurological deficits.
Time Frame: 48 hours post-ablation
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Groups:
- NAVISTAR® THERMOCOOL® (SNA Subpopulation Only): Version 3.0 of the Clinical Investigation Plan added a Subpopulation Neurological Assessments (SNA) designed to evaluate post-ablation generation of cerebral microemboli and associated neurological deficits.
  These assessments were done in a prospective, non-randomized manner, comparing subjects treated with the nMARQ system against control subjects treated with the NAVISTAR® THERMOCOOL® Irrigated Tip Catheter.
  Per study design, the data from the NAVISTAR® THERMOCOOL® subpopulation would be used for SNA analysis only. The data in this column are related for transparency; but cannot be compared statistically against the data from the Main Study group.
Arm/Group | nMARQ™ System (SNA Subpopulation) | NAVISTAR® THERMOCOOL® (SNA Subpopulation Only)
Number analyzed (Participants) | 19 | 17
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 Months post study procedure
Description: "Serious Adverse Events"/"Other (Not Including Serious) Adverse Events" tables: for the "NAVISTAR® THERMOCOOL® (SNA Subpopulation Only)" arm the "at Risk #" represents subjects enrolled and treated, including the 1 subject excluded from the SNA analysis due to missing neurological exams. (Excluding the subject not treated).
Groups:
- nMARQ™ System (Main Study): nMARQ™ is the Biosense Webster Pulmonary Vein Isolation System consists of Circular and Crescent Mapping and Ablation Catheters and the Multi-channel Radiofrequency Generator. This system is designed to facilitate electrophysiological mapping and transmit radiofrequency from multiple electrodes simultaneously for treating paroxysmal atrial fibrillation (PAF).
Arm/Group | nMARQ™ System (Main Study) | NAVISTAR® THERMOCOOL® (SNA Subpopulation Only)
Serious Adverse Events (participants affected / at risk) | 31/163 | 0/18
Other Adverse Events (participants affected / at risk) | 65/163 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nMARQ™ System (Main Study) (N=163) | NAVISTAR® THERMOCOOL® (SNA Subpopulation Only) (N=18)
Atrial flutter (Cardiac disorders) | 4 (6) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 4 (5) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 3 (3) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (2) | 0 (0)
Vessel puncture site haematoma (General disorders) | 2 (2) | 0 (0)
Arterial restenosis (Vascular disorders) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nMARQ™ System (Main Study) (N=163) | NAVISTAR® THERMOCOOL® (SNA Subpopulation Only) (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 8 (9) | 0 (0)
Atrial flutter (Cardiac disorders) | 4 (4) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 4 (4) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (4) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 5 (5) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 4 (6) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Allergic oedema (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 2 (2) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Polymerase chain reaction (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hemianopia homonymous (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.